CLINICAL TRIAL: NCT04448158
Title: Dynamics of Drug Resistance-associated Mutations in HIV-1 DNA Reverse Transcriptase Clearance During Effective Antiretroviral Therapy
Acronym: MUTARESERVOIR
Status: Completed | Type: Observational
Sponsor: Association de Recherche en Virologie et Dermatologie (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: ARVD-MUTARESERVOIR
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 5 years of virological suppression: - Patients harboring a fully suppressed HIV-1 plasma viral load for at least 5 years
  Interventions: Diagnostic Test: Genotypic Resistance Test
- 10 years of virological suppression: - Patients harboring a fully suppressed HIV-1 plasma viral load for at least 10 years
  Interventions: Diagnostic Test: Genotypic Resistance Test

INTERVENTIONS:
Diagnostic Test: Genotypic Resistance Test — A Genotypic Resistance Test by Sanger sequencing will be done after the period of virological suppression.
  * If M184V is still present no additional test will be performed.
  * If M184V is absent, we will go back in the previous samples (one per year) to determine the time point where the mutation has been cleared by sanger and UDS sequencing.

SUMMARY:
In view of the prolongation of patients living with HIV's life expectancy, the question of optimization of ART, which is still a life-long treatment, becomes central. While most patients achieve virological success, their treatments often need to be optimized in order to limit adverse events, drugs interactions and to improve adherence. The switch to dual regimen strategies represent one of the approaches for treatment optimization.

Circulating HIV-1 resistant variants can be archived in viral reservoirs, where they can persist for an unknown duration and reemerge in case of therapeutic selective pressure.

There is a need to assess the dynamic of archived Drug resistance associated mutations (DRAMs) clearance in cell-associated HIV DNA after a long period of virological control, in the perspective of ARVs recycling.

The investigators postulate that it could be interesting in the future to recycle ARV drugs (that where classified as "resistant" in the past) in subsequent regimen. The question is particularly important for 3TC/FTC for subsequent new regimen and for the use of dual regimen (disappearance of M184V).

Thus, the investigators propose a retrospective, longitudinal analysis on blood-cell-associated HIV-1 DNA samples in order to investigate by Sanger and Ultra Deep Sequencing the dynamics of decay and persistence of DNA HIV-1 variants harboring key drug resistance-associated mutations to NRTIs, in particular M184V, in patients with sustained virological control for at least 5 years under effective ART.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* Age ≥ 18 years
* Genotypic resistance test performed at time of failure and harboring at least M184V
* Fully suppressed HIV viral load for at least 5 or 10 years.
* Triple therapy or 2 drug regimen during the entire follow-up
* Availability of at least 1 stored whole blood sample /year

Exclusion Criteria:

* No genotypic resistance test available at time of failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The studied population will be composed of followed HIV infected patients of the center, of whom approximately 90% are under treatment and virologically suppressed, consecutively selected (in an anti-chronological order on the sample failure date) until gathering the requested number of patients meeting the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Detection of M184V mutation | One measure per year
  The persistence of M184V resistance mutation is defined by the detection of this mutation in 2 consecutive samples by Sanger and by a percentage of this mutation > 1% in 2 consecutive samples by UltraDeep Sequencing. The clearance of M184V is defined by the detection of this mutation by Sanger in a sample and the absence in the subsequent sample or a percentage of this mutation > 1% in a sample and a percentage < 1% in the subsequent sample.
Percentage of M184V mutation | One measure per year
  Percentage detected by UltraDeep Sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Geneviève MARCELIN, Principal Investigator — Sorbonne University; APHP
Locations (1):
- ARVD, Paris, France

IPD SHARING:
Plan to Share IPD: No